CLINICAL TRIAL: NCT01597947
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Intravenous (IV) ACHN-975 in Normal Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of ACHN-975 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Collaborators: Defense Medical Research and Development Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACHN-975-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ACHN-975

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: ACHN-975
- Arm B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ACHN-975 — Intravenous single dose
  Arms: Arm A
Drug: placebo — Intravenous single dose
  Arms: Arm B

SUMMARY:
This is a double-blind, randomized, placebo-controlled, single ascending dose study to assess the safety, tolerability, and PK of ACHN-975 in normal healthy volunteers. This study will take place in the US at one clinical site.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight between 40 and 100 kilograms (between ~88 pounds and ~220 pounds)
* Use of contraception
* Stable health
* Negative tests for alcohol, tobacco, and drugs of abuse

Key Exclusion Criteria:

* History of clinically significant disease
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Frequency of AEs | 7 days
Severity of AEs | 7 days

SECONDARY OUTCOMES:
Plasma concentrations of ACHN-975 | 2 days
Urine concentrations of ACHN-975 | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Achaogen, Inc.
Locations (1):
- Investigational Site, Durham, North Carolina, United States